CLINICAL TRIAL: NCT00494559
Title: Phase 4 Study of Pioglitazone on Neointima Volume and Inflammatory Markers in Diabetic Patients
Brief Title: The Effect of Pioglitazone on Neointima Volume and Inflammatory Markers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Principal Investigator, Soon Jun Hong, Associate professor, Korea University Anam Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRAISE
Record Dates: First submitted 2007-06-28; First posted 2007-06-29 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Diabetes Mellitus; Coronary Artery Stenosis
Keywords: Type 2 Diabetes; Pioglitazone; restenosis
MeSH Terms: conditions — Diabetes Mellitus; Coronary Stenosis; Diabetes Mellitus, Type 2 | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Actos (Experimental): Actos group: pioglitazone 15mg or 30mg
  Interventions: Drug: Pioglitazone
- Placebo (Placebo Comparator): Placebo group: placebo without active medication
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pioglitazone — Actos 15mg once a day before breakfast
  Other Names: Actos
  Arms: Actos
Drug: Placebo — Placebo drug with the same appearance as actos
  Arms: Placebo

SUMMARY:
People with diabetes mellitus are more prone to coronary heart disease, stroke, and peripheral vascular disease, and diabetes mellitus has been regarded as an independent risk factor for the progression of coronary artery disease. Several studies have been reported that diabetes increased the risk of cardiovascular mortality in both men and women. With the introduction of drug-eluting stents (DESs), the angiographic rates of restenosis at later months have reduced dramatically in several studies. However, even with DESs, diabetic patients showed increased rates of restenosis and late loss index compared with nondiabetic patients. Diabetes has been considered to be a predictor of poor prognosis after percutaneous coronary intervention with drug-eluting stents. Long-term clinical and angiographic outcomes after percutaneous coronary intervention (PCI) with drug-metal stents (DESs) have been demonstrated to be worse in diabetic patients compared with nondiabetic patients. In the era of DESs, no study has demonstrated the clinical and angiographic outcomes in diabetic patients after zotarolimus-eluting stent implantation by using intravascular ultrasound (IVUS).

Pioglitazone is used in the treatment of diabetic patients. Thiazolidinediones increase insulin sensitivity and show favorable effect on blood glucose levels and lipid profiles. The effect of pioglitazone on neointima volume and inflammatory markers has not been compared in prospective manner after zotarolimus-eluting stent implantation. The purpose of this prospective, randomized, single blinded trial is to compare the effect of pioglitazone on inflammatory markers and neointima volume by using IVUS in diabetic patients.

DETAILED DESCRIPTION:
With the introduction of the DES, the angiographic rates of restenosis have decreased dramatically but less prominently in diabetic patients. Even in the era of DES, diabetes remains a significant predictor of coronary restenosis especially in cases of small baseline and post PCI vessel size, longer stent length, current smokers, and high level of CRP. Restenosis remains a main clinical and angiographic concern after DES implantation especially in diabetic patients. Diabetes has been known as a major risk factor for in-stent restenosis after DES implantation.

1. Primary end point: Comparison of pioglitazone and placebo on 8 months follow-up neointima volume by intravascular ultrasound (IVUS).
2. Secondary end point: Comparison of pioglitazone and placebo on the changes in the levels of inflammatory markers (hsCRP, IL-6, TNF-α, adiponectin).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and above
* Gender eligible for study: both
* Diabetic patients either previously diagnosed or newly found diabetes.
* Fasting blood glucose ≥ 126 mg/dl or PP2 blood glucose ≥ 200 mg/dl for newly found diabetes.
* Patients with significant de novo coronary artery disease (diameter stenosis > 70%) requiring stent implantation (angina pectoris and/or exercise-induced ischemia).
* Patients with informed consent.

Exclusion Criteria:

* Acute ST-segment elevation myocardial infarction (MI)
* CTO lesions
* Left main lesions
* Diabetic patients with the use of thiazolidinediones within 3 months
* Previous history of PCI or bypass surgery
* Patients with any contraindications to the treatment of thiazolidinediones
* Pregnant or lactating patients
* Chronic alcohol or drug abuse
* Hepatic dysfunction
* Renal dysfunction
* Heart failure (EF < 50%)
* Expected life expectancy of < 1 year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Comparison of pioglitazone and placebo on 8 months follow-up neointima volume by intravascular ultrasound (IVUS). | 8 month follow-up

SECONDARY OUTCOMES:
Comparison of pioglitazone and placebo on the changes in the levels of inflammatory markers (hsCRP, IL-6, TNF-α, adiponectin). | 8 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Soon Jun Hong, MD, PhD, Principal Investigator — Korea University Anam Hospital; Sang Yup Lim, MD, PhD, Study Director — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea